CLINICAL TRIAL: NCT00784277
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, Parallel-Arm, Multicenter Study in Subjects With End-Stage Joint Disease to Compare the Frequency of Constipation Symptoms in SubjectsTreated With Tapentadol IR and Oxycodone IR Using a Bowel Function Patient Diary
Brief Title: A Study to Compare the Frequency of Constipation Symptoms With Tapentadol Immediate Release (IR) Treatment Versus Oxycodone IR Treatment in Patients With End-stage Joint Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Senior Director, Clinical Leader, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR014326; KF5503/41
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Results first posted 2012-02-13 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-01

CONDITIONS: Joint Diseases; Arthritis; Osteoarthritis
Keywords: Pain medication; Arthritis; Joint pain; Analgesia; Analgesics; tapentadol; CG5503; Nucynta
MeSH Terms: conditions — Joint Diseases; Arthritis; Osteoarthritis; Arthralgia; Agnosia | interventions — Tapentadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- 001 (Experimental): Tapentadol IR (CG5503) 50mg for 14 days
  Interventions: Drug: Tapentadol IR (CG5503)
- 002 (Experimental): Tapentadol IR (CG5503) 75mg for 14 days
  Interventions: Drug: Tapentadol IR (CG5503)
- 003 (Active Comparator): oxycodone IR 10mg for 14 days
  Interventions: Drug: oxycodone IR
- 004 (Placebo Comparator): placebo 1 capsule for 14 days
  Interventions: Drug: placebo
- 005 (Experimental): Tapentadol ER (CG5503) flexible dose tablets and capsules 2 x a day for 28 days (100-500mg/day)
  Interventions: Drug: Tapentadol ER (CG5503)
- 006 (Active Comparator): oxycodone CR flexible dose tablets and capsules 2 x a day for 28 days (20-60mg/day)
  Interventions: Drug: oxycodone CR
- 007 (Placebo Comparator): placebo Tablets and capsules 2 x a day for 28 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: oxycodone CR — flexible dose tablets and capsules 2 x a day for 28 days (20-60mg/day)
  Arms: 006
Drug: oxycodone IR — 10mg for 14 days
  Arms: 003
Drug: Tapentadol ER (CG5503) — flexible dose tablets and capsules 2 x a day for 28 days (100-500mg/day)
  Arms: 005
Drug: Tapentadol IR (CG5503) — 50mg for 14 days
  Arms: 001
Drug: Tapentadol IR (CG5503) — 75mg for 14 days
  Arms: 002
Drug: placebo — 1 capsule for 14 days
  Arms: 004
Drug: placebo — Tablets and capsules 2 x a day for 28 days
  Arms: 007

SUMMARY:
The purpose of this study is to compare bowel function/constipation that occurs during tapentadol treatment with that occuring during oxycodone treatment, as measured by the frequency of spontaneous bowel movements per week. The frequency of spontaneous bowel movements will be determined from a Bowel Function Patient Diary completed by the enrolled sujbects.

DETAILED DESCRIPTION:
Chronic pain from end-stage degenerative joint disease is often moderate to severe in intensity and results in a relatively constant level of pain requiring continuous pain relief medication. Despite available pain relief medications, 60% to 80% of subjects suffering from chronic pain are currently inadequately treated. Opioid pain medications are central to the effective treatment of moderate to severe pain. However, opioid therapy is frequently complicated by side effects. Constipation is one of the most commonly reported side effects and most debilitating. An opioid medication that provides pain relief with a reduced incidence of constipation symptoms would improve the capability of subjects to stay on medication to achieve the long-term relief they need. This is a randomized, double-blind, placebo- and active-controlled, parallel-arm, multicenter study with 4 treatment groups of subjects who have moderate to severe chronic pain from end-stage degenerative joint disease of the hip or knee and who are candidates for primary total or partial joint replacement. The study consists of 3 periods: a pretreatment period (a 14-day screening for study eligibility and a 7-day washout of any previously taken opioid medication), a double-blind treatment period (a 14-day IR treatment phase followed by a 28-day ER treatment phase), and a follow-up period (1 study-site visit within 4 days after the last dose of study drug is taken and 1 telephone contact within 10 to 14 days after the last dose of study drug is taken). On Day 1 of the IR treatment phase, patients will be randomly assigned to 1 of 4 possible treatment groups to receive 50 mg CG5503 IR, 75 mg CG5503 IR, 10 mg oxycodone IR, or placebo daily every 4 to 6 hours. At the beginning of the ER treatment phase, patients' study drugs will be transitioned to the ER form (by conversion from the IR to approximate equivalent total daily doses of the ER form) of their randomly assigned study drug of tapentadol ER, oxycodone CR, or placebo. The ER study drugs will be taken every 12 hours b.i.d. Dosages will be adjustable, with the study site personnel oversight, to ensure adequate pain relief is provided. Beginning with the washout period, patients will be given hand-held computer diaries in which to record their pain intensity, pain relief, bowel movement information, and answer questions on any nausea or vomiting that may occur. In addition, patients will write down the times and dosages of all medications they take during the study in a medication diary. Safety and tolerability will be assessed using physical examination, monitoring of adverse events, clinical and laboratory measures, and 12 lead ECG results. The first study hypothesis is that both tapentadol IR dosages are more effective than placebo in relieving pain based on the SPID score recorded by the patients over the first 5 days of the study. The second study hypothesis is that the Bowel Function Patient Diary results for both tapentadol IR dosages demonstrate improved tolerability compared to oxycodone IR 10 mg, based on the number of spontaneous bowel movements per week over the first 2 weeks of the study. In the IR treatment phase, each patient will take CG5503 IR 50 mg, CG5503 IR 75 mg, oxycodone IR 10 mg, or placebo orally every 4 to 6 hours for 14 days. In the ER treatment phase, dosages of the IR treatment groups will be converted to approximately equivalent dosages of the ER form of the assigned study drug: tapentadol ER, oxycodone CR, or placebo. Dosages may range from 100 to 500 mg/day of tapentadol ER and 20 to 60 mg/day of oxycodone CR taken orally 2x daily for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of osteoarthritis of the hip or knee
* End-stage degenerative joint disease
* Eligibility for primary unilateral total or partial joint replacement surgery
* Pain level moderate to severe and at such a level as to require daily doses of an opioid analgesic medication

Exclusion Criteria:

* Has a life-long history of seizure disorder or epilepsy
* Had any of the following within the preceding 1 year: mild or moderate traumatic brain injury, stroke, transient ischemic attack, or brain neoplasm
* Had a severe traumatic brain injury within 15 years of screening (consisting of one or more of the following: brain contusion, intracranial hematoma, either unconsciousness or post traumatic amnesia lasting for more than 24 hours)
* Joint pain not associated with gout, fibromyalgia, rheumatoid arthritis, other autoimmune disease
* History of alcohol or drug abuse
* chronic hepatitis B and C or HIV, active hepatitis B and C within 3 months
* Severely impaired renal function or moderately to severely impaired hepatic function
* History of cancer within past 2 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Etropolski M, Kelly K, Okamoto A, Rauschkolb C. Comparable efficacy and superior gastrointestinal tolerability (nausea, vomiting, constipation) of tapentadol compared with oxycodone hydrochloride. Adv Ther. 2011 May;28(5):401-17. doi: 10.1007/s12325-011-0018-0. Epub 2011 Apr 13. PMID 21494892

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1000 participants were screened, 598 were randomized, 596 participants received medication in the first part of the double-blind treatment period (IR treatment phase). A total of 463 participants received medication in the second part of the double-blind treatment period (ER treatment phase).
Groups:
- Placebo: IR Treatment : 1 capsule for 14 days
- Tapentadol 50 mg: IR Treatment : 50mg for 14 days
- Tapentadol 75 mg: IR Treatment : 75mg for 14 days
- Oxycodone: IR Treatment : 10mg for 14 days
- Placebo ER: ER Treatment : Tablets and capsules 2 x a day for 28 days
- Tapentadol ER: ER Treatment : flexible dose tablets and capsules 2 x a day for 28 days (100-500mg/day)
- Oxycodone CR: ER Treatment : flexible dose tablets and capsules 2 x a day for 28 days (20-60mg/day)
Period: IR Treatment
Arm/Group | Placebo | Tapentadol 50 mg | Tapentadol 75 mg | Oxycodone | Placebo ER | Tapentadol ER | Oxycodone CR
Started | 148 | 151 | 154 | 143 | 0 ("0" in ER column indicates this reporting group is not relevant to IR phase.) | 0 ("0" in ER column indicates this reporting group is not relevant to IR phase.) | 0 ("0" in ER column indicates this reporting group is not relevant to IR phase.)
Completed | 132 | 134 | 126 | 100 | 0 | 0 | 0
Not Completed | 16 | 17 | 28 | 43 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 8 | 19 | 35 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 4 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 4 | 6 | 0 | 0 | 0
Not completed — Resolution Of Pain | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 3 | 3 | 2 | 0 | 0 | 0
Period: ER Treatment
Arm/Group | Placebo | Tapentadol 50 mg | Tapentadol 75 mg | Oxycodone | Placebo ER | Tapentadol ER | Oxycodone CR
Started | 0 ("0" in IR column indicates this reporting group is not relevant to ER phase.) | 0 ("0" in IR column indicates this reporting group is not relevant to ER phase.) | 0 ("0" in IR column indicates this reporting group is not relevant to ER phase.) | 0 ("0" in IR column indicates this reporting group is not relevant to ER phase.) | 122 (10 participants who had completed IR treatment have not taken any ER treatment.) | 250 (10 participants who had completed IR treatment have not taken any ER treatment.) | 91 (9 participants who had completed IR treatment have not taken any ER treatment.)
Completed | 0 | 0 | 0 | 0 | 113 | 226 | 76
Not Completed | 0 | 0 | 0 | 0 | 9 | 24 | 15
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 7 | 7
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 3 | 4 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 5 | 3
Not completed — Study Medication Non-Compliant | 0 | 0 | 0 | 0 | 2 | 3 | 3
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Tapentadol 50 mg: IR Treatment : 50mg capsule for 14 days
- Tapentadol 75 mg: IR Treatment : 75mg capsule for 14 days
- Oxycodone: IR Treatment : 10mg capsule for 14 days
- Total: Total of all reporting groups
Arm/Group | Placebo | Tapentadol 50 mg | Tapentadol 75 mg | Oxycodone | Total
Number analyzed (Participants) | 148 | 151 | 154 | 143 | 596
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 110 | 113 | 114 | 109 | 446
  >=65 years | 38 | 38 | 40 | 34 | 150
Age Continuous [Mean (Standard Deviation); unit: years] | 58.8 (9.57) | 58 (9.47) | 58.4 (7.66) | 59.4 (7.94) | 58.7 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 93 | 75 | 81 | 349
  Male | 48 | 58 | 79 | 62 | 247
Region Enroll [Number; unit: Participants]
  Canada | 32 | 36 | 37 | 34 | 139
  USA | 116 | 115 | 117 | 109 | 457

OUTCOME MEASURES:

1. Primary Outcome: 5-Day Sum of Pain Intensity Difference (SPID5)
Description: SPID5 was calculated as the weighted (weights is taken as the number of hours elapsed since the previous measurement) sum of the PID collected up to 5 days. Pain intensity (PI) score is calculated as the average PI over the past 12 hours using an 11-point (0 to 10) numerical rating scale (NRS) where "0" is no pain and "10" is pain as bad as you can imagine. The difference between baseline PI at the qualifying period and current PI is pain intensity difference (PID).
Time Frame: Day 1 to Day 5
Population: Intention To Treat (ITT) population : One participant who has been treated is not included in the ITT population as no baseline pain assessment was available (Arm: Tapentadol 50 mg).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Tapentadol 50 mg | Tapentadol 75 mg | Oxycodone
Number analyzed (Participants) | 148 | 150 | 154 | 143
Units on a scale | 98.6 (134.73) | 153.1 (184.07) | 161.8 (187.31) | 218.4 (208.64)
Statistical Analysis 1: Comparison: Placebo vs Tapentadol 50 mg; Test type: Superiority or Other; p = 0.007, ANCOVA — P-value is adjusted for multiplicity for comparison against placebo using Hochberg's test; The model includes treatment and pooled center as factors and baseline pain intensity score as covariate; Difference in Least-Squares Means = 55.1, 95% CI [15.11 to 95.13], Standard Error of Mean 20.37 — The 95% confidence interval is unadjusted for multiplicity
Statistical Analysis 2: Comparison: Placebo vs Tapentadol 75 mg; Test type: Superiority or Other; p = 0.004, ANCOVA — P-value is adjusted for multiplicity for comparison against placebo using Hochberg's test; The model includes treatment and pooled center as factors and baseline pain intensity score as covariate; Difference in Least-Squares Means = 63.4, 95% CI [23.67 to 103.13], Standard Error of Mean 20.23 — The 95% confidence interval is unadjusted for multiplicity

2. Primary Outcome: Spontaneous Bowel Movements Per Week (SBMs/Week)
Description: The number of SBM over the 14-day IR treatment phase was determined from the Bowel Function Patient Diary and factored to enable a per week value to be used. An SBM is defined as any BM that has occurred without the use of a laxative, enema, suppository, or manual manipulation within the previous 24 hours.
Time Frame: Week 1 to Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of stools/week
Arm/Group | Placebo | Tapentadol 50 mg | Tapentadol 75 mg | Oxycodone
Number analyzed (Participants) | 148 | 150 | 154 | 143
number of stools/week | 9.9 (5.16) | 9.0 (4.04) | 8.6 (4.65) | 6.7 (5.44)
Statistical Analysis 1: Comparison: Placebo vs Oxycodone; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is adjusted for multiplicity for comparison against Oxycodone using Hochberg's test; The model includes treatment and pooled center as factors and baseline value as covariate; Difference in Least-Squares Means = 3.1, 95% CI [2.22 to 4.01], Standard Error of Mean 0.46 — The 95% confidence interval is unadjusted for multiplicity
Statistical Analysis 2: Comparison: Tapentadol 50 mg vs Oxycodone; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is adjusted for multiplicity for comparison against Oxycodone using Hochberg's test; The model includes treatment and pooled center as factors and baseline value as covariate; Difference in Least-Squares Means = 2.2, 95% CI [1.34 to 3.12], Standard Error of Mean 0.45 — The 95% confidence interval is unadjusted for multiplicity
Statistical Analysis 3: Comparison: Tapentadol 75 mg vs Oxycodone; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is adjusted for multiplicity for comparison against Oxycodone using Hochberg's test; The model includes treatment and pooled center as factors and baseline value as covariate; Difference in Least-Squares Means = 1.6, 95% CI [0.72 to 2.50], Standard Error of Mean 0.45 — The 95% confidence interval is unadjusted for multiplicity

ADVERSE EVENTS:
Description: Only participants who had at least one of the TEAEs listed in the Other (non Serious) AE table are included in the Total no. participants with Non-Serious Adverse Events.
Arm/Group | Placebo | Tapentadol 50 mg | Tapentadol 75 mg | Oxycodone | Placebo ER | Tapentadol ER | Oxycodone CR
Serious Adverse Events (participants affected / at risk) | 1/148 | 1/151 | 0/154 | 1/143 | 0/122 | 1/250 | 0/91
Other Adverse Events (participants affected / at risk) | 48/148 | 65/151 | 88/154 | 98/143 | 23/122 | 80/250 | 36/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=148) | Tapentadol 50 mg (N=151) | Tapentadol 75 mg (N=154) | Oxycodone (N=143) | Placebo ER (N=122) | Tapentadol ER (N=250) | Oxycodone CR (N=91)
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=148) | Tapentadol 50 mg (N=151) | Tapentadol 75 mg (N=154) | Oxycodone (N=143) | Placebo ER (N=122) | Tapentadol ER (N=250) | Oxycodone CR (N=91)
Nausea (Gastrointestinal disorders) | 11 | 26 | 31 | 57 | 5 | 23 | 12
Constipation (Gastrointestinal disorders) | 22 | 21 | 28 | 42 | 10 | 37 | 18
Vomiting (Gastrointestinal disorders) | 1 | 7 | 13 | 34 | 5 | 13 | 6
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 7 | 5 | 5 | 13 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 4 | 9 | 6 | 1 | 3 | 1
Somnolence (Nervous system disorders) | 5 | 20 | 14 | 17 | 2 | 8 | 2
Dizziness (Nervous system disorders) | 6 | 17 | 35 | 25 | 4 | 5 | 3
Headache (Nervous system disorders) | 12 | 6 | 7 | 15 | 7 | 8 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 4 | 13 | 0 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less